CLINICAL TRIAL: NCT04511130
Title: A Phase 2 Study of Donor-Derived Multi-Tumor-Associated Antigen Specific T Cells (MT-401) Administered to Patients With Acute Myeloid Leukemia (AML) Following Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of MT-401 in Patients With AML Following Stem Cell Transplant
Acronym: ARTEMIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite a plan to enroll ~195-210 participants, the ARTEMIS study was closed due to the long vein-to-vein manufacturing timeline of MT-401 after 38 participants received the autologous MT-401.
Sponsor: Marker Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MRKR-19-401; FD-R-7272 (Other Grant/Funding Number: Office of Orphan Products Development)
Record Dates: First submitted 2020-07-30; First posted 2020-08-13 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MT-401 following HSCT (Experimental): Treatment with MT-401 at 90 days following HSCT
  Interventions: Drug: MT-401
- Standard of Care following HSCT (No Intervention): Standard of Care
- MT-401 following relapse (Experimental): Treatment with MT-401 following relapse after first HSCT
  Interventions: Drug: MT-401

INTERVENTIONS:
Drug: MT-401 — MT-401 (zedenoleucel) is an allogeneic multi-tumor-associated antigen (MultiTAA)-specific T cell product manufactured under Good Manufacturing Practice (GMP) using donor-derived T cells obtained from apheresis.
  Other Names: zedenoleucel
  Arms: MT-401 following HSCT; MT-401 following relapse

SUMMARY:
This study is a Phase 2 multicenter study with a Safety Lead-in evaluating safety and efficacy of MT-401 administration to patients with AML, who have received their first allogeneic HSCT. The dose administered is 50 x 10^6 cells (flat dosing).

DETAILED DESCRIPTION:
This study is in patients aged ≥18 years old undergoing or having relapsed after their first allogeneic HSCT (matched sibling, matched unrelated donor, or haploidentical transplants) for AML.

Potential patients for the study may be screened/enrolled:

• Prior to their first allogeneic HSCT.

or

• Patients experiencing their first relapse post-allogeneic transplant.

Patients eligible for the study will be placed into one of two groups:

* Adjuvant (Group 1): Patients screened prior to their HSCT with CR without minimal residual disease (CRMRD-) at 85-130 days post transplant will be randomized (1:1) in an unblinded fashion to:

  * MT-401 (Arm A)
  * SOC (Arm B)
* Active Disease: (Group 2): Patients meeting the following criteria will be assigned to Group 2 and will receive MT 401:

  * Patients who experience relapse (patients with MRD [MRD+] or frank relapse) at or prior to post-transplant Day 85-130
  * Patients in Arm B of Group 1 (SOC) who develop relapse (MRD+ or frank relapse) post-HSCT (crossover patients)
  * Patients who do not consent prior to HSCT but are experiencing their first relapse (MRD+ or frank relapse) and have the same donor available for manufacturing

ELIGIBILITY:
Inclusion Criteria

1. First allogeneic HSCT, in ≤ CR2, and MRD negative prior to transplant (including matched sibling, MUD with at least 6 of 8 HLA markers, or haploidentical with at least 5 of 10 HLA markers) as:

   * Adjuvant therapy for AML (Group 1) at 85-130 days post-HSCT defined as patients with CRMRD; or
   * Treatment for refractory/relapsed AML (first relapse post-HSCT) when disease occurs after transplant (Group 2) defined as

     * First relapse (MRD+ or frank relapse) post-HSCT
     * Patients in Arm 1B (SOC) who experience first relapse (MRD+ or frank relapse) post HSCT
   * Safety Lead-in defined as patients who fit all the criteria for Group 2 only
2. Are ≥18 years of age
3. Karnofsky/ Lansky score of ≥60
4. Life expectancy ≥12 weeks
5. Adequate blood, liver, and renal function

   * Blood: Hemoglobin ≥7.0 g/dL (can be transfused)
   * Liver: Bilirubin ≤2X upper limit of normal; aspartate aminotransferase ≤3X upper limit of normal
   * Renal: Serum creatinine ≤2X upper limit of normal or measured or calculated creatinine clearance ≥45mL/min

7. Patients are allowed to be on experimental conditioning regimens prior to transplant if no planned maintenance therapy post-transplant.

8. In Group 2, patients may receive bridging therapy at the investigators' discretion in situations where MT-401 is not ready for administration or the treating physician believes the patient would benefit

Exclusion Criteria

1. Clinically significant or severely symptomatic intercurrent infection
2. Pregnant or lactating
3. For Group 1, anti-neoplastic therapy after HSCT and prior to or during dosing of MT-401
4. For Group 2, concomitant anti-neoplastic therapy during or after dosing of MT-401
5. Evidence of acute or chronic GVHD ≥Grade 2 (exception: acute or chronic Grade 2 GVHD of skin allowed if stable) within one week prior to receiving MT-401

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Safety Lead-In | Baseline through Cycle 1 (28 Days)
  Number of participants with MT-401 Dose Limiting Toxicities (DLTs)
Phase 2 Adjuvant Group | Up to 24 months after the first participant is randomized
  Relapse Free Survival (RFS), defined as the time from randomization to first disease recurrence or death from any cause.
Phase 2 Active Disease Group | Up to 12 months
  Complete Remission (CR), per European LeukemiaNet (ELN) 2017 criteria
Phase 2 Active Disease Group | Up to 24 months
  Duration of CR (DOCR), defined as the time from the first observation of CR through disease recurrence or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Nishan Rajakumaraswamy, MD, Study Director — Marker Therapeutics
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Moores Cancer Center at University of Californa San Diego, La Jolla, California
  - UCLA Department of Medicine, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinical Cancer Center-Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mayo Clinic Cancer Center-Rochester, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack UMC, Hackensack, New Jersey
  - Weill Cornell Medicine | NewYork-Presbyterian, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT04511130/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT04511130/SAP_001.pdf